CLINICAL TRIAL: NCT03194542
Title: A Phase-2 Study To Determine Efficacy and Safety of Luspatercept in Subjects With Myeloproliferative Neoplasm-Associated Myelofibrosis and Anemia With or Without Red Blood Cell-Transfusion Dependence
Brief Title: A Safety and Efficacy Study to Evaluate Luspatercept in Subjects With Myeloproliferative Neoplasm-associated Myelofibrosis Who Have Anemia With and Without Red Blood Cell-transfusion Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACE-536-MF-001; 2017-000322-35 (EudraCT Number); U1111-1197-1202 (Registry Identifier: WHO)
Record Dates: First submitted 2017-06-15; First posted 2017-06-21 (Actual); Results first posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Primary Myelofibrosis; Anemia
Keywords: Luspatercept; ACE-536; Myeloproliferative Neoplasm-Associated Myelofibrosis; Primary Myelofibrosis; Post-Polycythemia Vera Myelofibrosis; Post-Essential Thrombocythemia; Anemia; Red Blood Cell (RBC) Transfusion; Ruxolitinib
MeSH Terms: conditions — Primary Myelofibrosis; Anemia | interventions — luspatercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Luspatercept in subjects with MPN-associated myelofibrosis (Experimental): Subjects across each of the cohorts (Cohort 1, Cohort 2, Cohort 3A, and Cohort 3B) will receive luspatercept.
  Interventions: Drug: Luspatercept

INTERVENTIONS:
Drug: Luspatercept — Luspatercept is a recombinant fusion protein consisting of a modified form of the extracellular domain of the human active in receptor type IIB linked to the IgG1 Fc domain. Luspatercept, through a mechanism of action different from erythropoietin, works to correct ineffective erythropoiesis by promoting late-stage maturation of erythroblasts.
  Other Names: ACE-536

SUMMARY:
This is a Phase 2, multicenter, open-label study to evaluate the efficacy and safety of luspatercept in subjects with MPN-associated myelofibrosis and anemia with and without RBC-transfusion dependence. The study is divided into a Screening Period, a Treatment Period (consisting of a Primary Phase, a Day 169 Disease Response Assessment, and an Extension Phase), followed by a Posttreatment Follow-up Period.

DETAILED DESCRIPTION:
Subjects satisfying the eligibility criteria will be assigned to 1 of the following cohorts (which are enrolling in parallel) based on their eligibility:

* Cohort 1 (subjects with anemia only that are not currently receiving RBC transfusions) - Cohort 2: (subjects that are RBC-transfusion dependent)
* Cohort 3A: (subjects on ruxolitinib as part of their standard of care therapy that have anemia only)
* Cohort 3B: (subjects on ruxolitinib as part of their standard of care therapy that are RBC-transfusion dependent) Overall, the study will enroll approximately 100 subjects worldwide.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study (with the enrollment date defined as the date in which the subject is assigned a cohort in Integrated Response Technology [IRT]) and receive their first dose of luspatercept:

1. Subject is ≥18 years of age at the time of signing the informed consent form (ICF).
2. Subject has Myeloproliferative neoplasm (MPN)-associated myelofibrosis (PMF, post- Post-polycythemia vera myelofibrosis (PV MF), and/or Post-essential thrombocythemia myelofibrosis (post-ET MF)) as confirmed from the most recent local bone marrow biopsy report according to the World Health Organization 2016 criteria.
3. Subject has anemia defined as:

   1. Cohorts 1 and 3A

      * Obtain ≥ 3 Hemoglobin (Hgb) levels of ≤ 9.5 g/dL recorded on ≥ 3 different days, including the day of dosing, in the 84-day period immediately up to the C1D1 date. There must be ≥ 14 days in between each Hgb measurement. No subjects with an interval ≥ 42 days between hemoglobin measurements will be enrolled.
      * There must not be any Red blood cell (RBC) transfusions within the 84-day period immediately up to the C1D1 date.
   2. Cohorts 2 and 3B

      * Average RBC-transfusion frequency: 4 to 12 RBC units/84 days immediately up to the C1D1 date. There must be no interval > 56 days without ≥ 1 RBC-transfusion.
      * Subjects must have a Hgb value of < 13 g/dL on C1D1 prior to luspatercept administration.
      * Only RBC transfusions given when the Hgb ≤ 9.5 g/dL are scored in determining eligibility.
4. Subject has an Eastern Cooperative Oncology Group (ECOG) performance score of ≤ 2.
5. Subject is not anticipated during the 6 months from the C1D1 date to receive a hematopoietic cell transplant.
6. A female of childbearing potential (FCBP) for this study is defined as a female who: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (ie, has had menses at any time in the preceding 24 consecutive months). FCBP participating in the study must:

   1. Have 2 negative pregnancy tests as verified by the Investigator prior to starting study therapy. She must agree to ongoing pregnancy testing during the course of the study, and after end of study treatment. This applies even if the subject practices true abstinence* from heterosexual contact.
   2. Either commit to true abstinence* from heterosexual contact (which must be reviewed on a monthly basis and source documented) or agree to use, and be able to comply with, effective contraception** without interruption, 28 days prior to starting investigational product, during the study therapy (including dose interruptions), and for 12 weeks (approximately 5 times the mean terminal halflife of luspatercept based on multiple-dose pharmacokinetics [PK] data) after discontinuation of study therapy.
7. Male subjects must:

   a. Practice true abstinence (which must be reviewed on a monthly basis) or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for at least 12 weeks (approximately 5 times the mean terminal half-life of luspatercept based on multiple-dose PK data) following investigational product discontinuation, even if he has undergone a successful vasectomy
8. Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
9. Subject is willing and able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment (with the enrollment date defined as the date in which the subject is assigned a cohort in Integrated Response Technology (IRT)):

1. Subject use of hydroxyurea or other drugs with potential effects on hematopoiesis or ongoing adverse events from previous treatment ≤ 112 days immediately up to the enrollment date.

   a. Systemic corticosteroids are permitted for nonhematological conditions providing the subject is receiving a stable or decreasing dose for ≥ 84 days immediately up to enrollment and is receiving a constant dose equivalent to ≤ 10 mg prednisone for the 28 days immediately up to enrollment.
2. Cohort 1 and 2 only: subjects treated with Janus kinase 2 gene (JAK2) inhibitors ≤ 112 days immediately up to the enrollment date or if anticipated/substantial likelihood for subject to receive ruxolitinib within the first 168 days on the study.
3. Cohort 3 only: subjects not receiving ruxolitinib:

   1. for at least 280 days (40 weeks) without interruptions exceeding 2 consecutive weeks
   2. on a stable daily dose for at least 112 days (16 weeks) immediately up to the enrollment date as part of their standard-of-care therapy.
4. Subject use of ESAs or androgenic steroids ≤ 112 days immediately up to the enrollment date.
5. Initiation of iron chelation therapy (ICT) or change with ICT dose within ≤ 112 days up to the enrollment date.
6. Subject with anemia from iron deficiency, B12 and folate deficiencies, hemolytic anemia, infection, or bleeding.
7. Pregnant or breastfeeding females.
8. Subject with blood myeloblasts ≥ 5%.
9. Subject with major surgery within 8 weeks up to the enrollment date. Subject must have completely recovered from any previous surgery immediately up to the enrollment date.
10. Subject with prior history of malignancies, other than disease under study, unless the subject has been free of the disease for ≥ 5 years. However, subject with the following history/concurrent conditions is allowed:

    * Basal or squamous cell carcinoma of the skin
    * Carcinoma in situ of the cervix
    * Carcinoma in situ of the breast
    * Incidental histologic finding of prostate cancer (T1a or T1b using the tumor, nodes, metastasis [TNM] clinical staging system)
11. Subject with prior therapy of luspatercept or sotatercept.
12. Subject participation in any other clinical protocol or investigational trial that involves administration of experimental therapy and/or therapeutic devices within 30 days immediately up to the enrollment date.
13. Subject with prior hematopoietic cell transplant.
14. Subject with any of the following laboratory abnormalities:

    * Neutrophils < 1 x 109/L
    * White blood count (WBC) > 100 x 109/L
    * Platelets

      * Cohorts 1 and 2: < 25 x 109/L
      * Cohort 3A and 3B: < 50 x 109/L
      * All Cohorts: > 1000 x 109/L
    * Estimated glomerular filtration rate < 45 mL/min/1.73 m2 (via the 4-variable modification of diet in renal disease [Modification of diet in renal disease (MDRD)] formula)
    * Aspartate aminotransferase (AST) or alanine transaminase (ALT) > 3.0 x upper limit of normal (ULN)
    * Direct bilirubin ≥ 2 x ULN

      * higher levels are acceptable if these can be attributed to active red blood cell precursor destruction within the bone marrow (ie, ineffective erythropoiesis)
    * Uncontrolled hyperthyroidism or hypothyroidism
15. Subject with stroke, deep venous thrombosis, pulmonary or arterial embolism within 6 months immediately up to the enrollment date.
16. Subject with diastolic blood pressure ≥ 90 mmHg or systolic blood pressure ≥ 140 mmHg measured during the Screening Period despite appropriate treatment.
17. Subject with inadequately controlled heart disease and/or have a known left ventricular ejection fraction <35%.
18. Subject with history of severe allergic or anaphylactic reactions or hypersensitivity to recombinant proteins or excipients in the investigational product (see luspatercept Investigator's Brochure (IB)).
19. Subject with uncontrolled systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment).
20. Subject with human immunodeficiency virus (HIV), evidence of active infectious Hepatitis B (HepB), and/or evidence of active Hepatitis C (HepC).
21. Subject with any significant medical condition, laboratory abnormality, psychiatric illness, or is considered vulnerable by local regulations (eg, imprisoned or institutionalized) that would prevent the subject from participating in the study.
22. Subject with any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
23. Subject with any condition or concomitant medication that confounds the ability to interpret data from the study.
24. Subject on anticoagulant therapy not under appropriate control or subject not on a stable dose of anticoagulant therapy for ≥ 8 weeks up to the enrollment date.
25. Subject on anagrelide within 28 days immediately up to the enrollment date.
26. Subject with a major bleeding event (defined as symptomatic bleeding in a critical area or organ and/or bleeding causing a decrease in hemoglobin of ≥ 2g/dL or leading to transfusion of ≥ 2 units of packed red cells) in the last 6 months prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (47):
- United States (20):
  - Local Institution - 102, Phoenix, Arizona
  - Mayo Clinic - Arizona, Phoenix, Arizona
  - Local Institution - 103, Stanford, California
  - Stanford Cancer Center, Stanford, California
  - Local Institution - 101, Jacksonville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Local Institution - 107, Orange City, Florida
  - Mid Florida Hematology and Oncology Centers, PA, Orange City, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Local Institution - 108, Tampa, Florida
  - Local Institution - 104, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Local Institution - 109, Cleveland, Ohio
  - Avera Research Institute, Sioux Falls, South Dakota
  - Local Institution - 105, Sioux Falls, South Dakota
  - Local Institution - 100, Houston, Texas
  - MD Anderson Cancer Center The University of Texas, Houston, Texas
  - Local Institution - 106, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
- France (8):
  - CHRU de Brest - Hopital Morvan, Brest
  - Local Institution - 203, Brest
  - Centre Hospitalier de Lens, Lens
  - Local Institution - 201, Lens
  - Hopital Saint Louis, Paris
  - Local Institution - 200, Paris
  - Gustave Roussy, Villejuif
  - Local Institution - 202, Villejuif
- Italy (10):
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Local Institution - 304, Bergamo
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Local Institution - 300, Florence
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Local Institution - 301, Pavia
  - Istituto Clinico Humanitas, Rozzano (MI)
  - Local Institution - 303, Rozzano (MI)
  - Local Institution - 302, Varese
  - Ospedale di Circolo di Varese, Varese
- United Kingdom (9):
  - Belfast Health and Social Care Trust, Belfast Northern Ireland
  - Local Institution - 404, Cardiff
  - University Hospital of Wales, Cardiff
  - Local Institution - 400, Headington, Oxford
  - University of Oxford, Headington, Oxford
  - Guy's and St Thomas' NHS Foundation Trust - Guy's Hospital, London
  - Local Institution - 403, London
  - Imperial College London, London
  - Local Institution - 402, London

REFERENCES:
- [Derived] Gerds AT, Harrison C, Kiladjian JJ, Mesa R, Vannucchi AM, Komrokji R, Bose P, Kremyanskaya M, Mead AJ, Gotlib J, Rose S, Sanabria F, Marsousi N, Giuseppi AC, Jiang H, Palmer JM, McCaul K, Ribrag V, Passamonti F. Safety and efficacy of luspatercept for the treatment of anemia in patients with myelofibrosis. Blood Adv. 2024 Sep 10;8(17):4511-4522. doi: 10.1182/bloodadvances.2024012939. PMID 38820422
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Anemia Only; Cohort 2: RBC-Transfusion Dependent: Participants receive a starting dose level of luspatercept at 1.0 mg/kg subcutaneous injection every 3 weeks (administered on Day 1 of each 21-day treatment cycle). The starting dose can be titrated (increased) during the Treatment Period to 1.33 mg/kg, up to a maximum of 1.75 mg/kg, provided that the participant meets the appropriate criteria. The participant's dose may also be delayed, reduced, or discontinued, depending on the specific criteria.
- Cohort 3A: Anemia Only (Stable Dose of Ruxolitinib); Cohort 3B: RBC-Transfusion Dependent (Stable Dose of Ruxolitinib): Participants receive a starting dose level of luspatercept at 1.0 mg/kg subcutaneous injection every 3 weeks (administered on Day 1 of each 21-day treatment cycle) while being on a stable dose of ruxolitinib for at least 112 days immediately prior to the enrollment date. The starting dose can be titrated (increased) during the Treatment Period to 1.33 mg/kg, up to a maximum of 1.75 mg/kg, provided that the participant meets the appropriate criteria. The participant's dose may also be delayed, reduced, or discontinued, depending on the specific criteria.
Period: Overall Study
Arm/Group | Cohort 1: Anemia Only | Cohort 2: RBC-Transfusion Dependent | Cohort 3A: Anemia Only (Stable Dose of Ruxolitinib) | Cohort 3B: RBC-Transfusion Dependent (Stable Dose of Ruxolitinib)
Started | 22 | 21 | 14 | 38
Completed (Treatment ongoing) | 0 | 0 | 0 | 0
Not Completed | 22 | 21 | 14 | 38
Not completed — Participant to Receive Bone Marrow Transplant | 1 | 0 | 0 | 0
Not completed — Rollover to Long-term follow-up Protocol | 1 | 1 | 0 | 5
Not completed — Per Protocol Repeat Blasts of 10% | 1 | 0 | 1 | 0
Not completed — Loss of Response | 4 | 2 | 3 | 4
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 2 | 2 | 2 | 6
Not completed — Withdrawal by Subject | 2 | 1 | 5 | 4
Not completed — Progressive Disease | 1 | 0 | 1 | 1
Not completed — Adverse Event | 1 | 2 | 0 | 5
Not completed — Death | 1 | 2 | 0 | 5
Not completed — Completed the primary treatment phase but did not meet clinical benefit criteria | 8 | 10 | 2 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Anemia Only | Cohort 2: RBC-Transfusion Dependent | Cohort 3A: Anemia Only (Stable Dose of Ruxolitinib) | Cohort 3B: RBC-Transfusion Dependent (Stable Dose of Ruxolitinib) | Total
Number analyzed (Participants) | 22 | 21 | 14 | 38 | 95
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69 (8.87) | 73.9 (5.71) | 65.4 (8.45) | 71.3 (5.80) | 70.5 (7.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 7 | 15 | 37
  Male | 13 | 15 | 7 | 23 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 1 | 3
  Not Hispanic or Latino | 16 | 19 | 14 | 32 | 81
  Unknown or Not Reported | 4 | 2 | 0 | 5 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 3 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 2 | 3
  White | 16 | 18 | 10 | 30 | 74
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 0 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Anemia Responses Over Any 84-Day Period During the Primary Treatment Period
Description: The number of participants that achieved anemia response as it relates to hemoglobin (Hgb) increase and red blood cell (RBC)-transfusion independence is defined below:
  Cohorts 1 (anemia only) and 3A: The number of participants achieving ≥ 1.5 g/dL hemoglobin increase from baseline over any consecutive 84-day period without an RBC transfusion from Day 1 up through and including Day 168.
  Cohorts 2 (RBC-transfusion dependent) and 3B: The number of participants who become RBC-transfusion free over any consecutive 84-day period from Day 1 up through and including Day 168.
  Baseline value is defined as the last value (including "unscheduled") measured on or before the first dose.
Time Frame: Any consecutive "rolling" 84-day period from Day 1 through and including Day 168
Population: Intent-to-treat (ITT) population: All enrolled participants regardless of whether or not the participant received luspatercept.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Anemia Only | Cohort 2: RBC-Transfusion Dependent | Cohort 3A: Anemia Only (Stable Dose of Ruxolitinib) | Cohort 3B: RBC-Transfusion Dependent (Stable Dose of Ruxolitinib)
Number analyzed (Participants) | 22 | 21 | 14 | 38
Participants | 3 | 2 | 2 | 10

2. Secondary Outcome: Time to Anemia Response During the Primary Treatment Period
Description: Time to anemia response follows the definitions below:
  Cohorts 1 (anemia only) and 3A: Time between first administration of luspatercept and the first hemoglobin increase of ≥ 1.5 g/dL from baseline that starts a consecutive 84-day period of consecutive increase ≥ 1.5 g/dL without RBC transfusions.
  Cohorts 2 (RBC-transfusion dependent) and 3B: Time between first administration of luspatercept and the first day of an RBC transfusion-free period of 84 days.
  Baseline value is defined as the last value (including "unscheduled") measured on or before the first dose.
Time Frame: From first dose up to first onset of anemia response (calculated from Day 1 through and including Day 168)
Population: ITT population who achieved anemia response. (Intent-to-treat (ITT) population: All enrolled participants regardless of whether or not the participant received luspatercept.)
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Cohort 1: Anemia Only | Cohort 2: RBC-Transfusion Dependent | Cohort 3A: Anemia Only (Stable Dose of Ruxolitinib) | Cohort 3B: RBC-Transfusion Dependent (Stable Dose of Ruxolitinib)
Number analyzed (Participants) | 3 | 2 | 2 | 10
Days | 57.3 (14.36) | 2.0 (0.00) | 63.5 (30.41) | 30.7 (27.22)

3. Secondary Outcome: Duration of Anemia Response
Description: The duration of anemia response is defined as the duration of time from first day of longest response to the last day of longest response. Participants who achieved and maintained the anemia response at the time of the analysis are censored at the efficacy cutoff date. For Cohorts 1 and 3A, an anemia responder was defined as a subject with ≥ 1.5 g/dL hemoglobin increase from baseline over any consecutive 84-day period without an RBC transfusion. For Cohorts 2 and 3B, an anemia responder was defined as a subject who becomes RBC transfusion free over any consecutive 84-day period.
  Baseline value is defined as the last value (including "unscheduled") measured on or before the first dose.
Time Frame: From first dose through last day of longest response (calculated from Day 1 through end of treatment, up to approximately 232 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Cohort 1: Anemia Only | Cohort 2: RBC-Transfusion Dependent | Cohort 3A: Anemia Only (Stable Dose of Ruxolitinib) | Cohort 3B: RBC-Transfusion Dependent (Stable Dose of Ruxolitinib)
Number analyzed (Participants) | 3 | 2 | 2 | 10
Days | 457.7 (611.20) | 623.0 (29.70) | 88.5 (6.36) | 534.7 (527.67)

4. Secondary Outcome: The Number of RBC Units Transfused Per Participant Per 28 Days (Cohorts 2 and 3B Only)
Description: Frequency of RBC transfusion is defined as the mean number of RBC units transfused per participant every 4 weeks (28 days). The primary treatment period is from Day 1 to and including Day 168. The entire treatment period is from Day 1 through the end of treatment.
Time Frame: From Day 1 through end of treatment (up to approximately 232 weeks).
Population: Intent-to-treat (ITT) population: All enrolled participants regardless of whether or not the participant received luspatercept. Pre-specified to be collected for Cohorts 2 and 3B only.
Measure: Mean (Standard Deviation); unit: RBC Units
Arm/Group | Cohort 2: RBC-Transfusion Dependent | Cohort 3B: RBC-Transfusion Dependent (Stable Dose of Ruxolitinib)
Number analyzed (Participants) | 21 | 38
RBC Units
  Primary Treatment Period | 2.76 (1.967) | 1.49 (1.345)
  Entire Treatment Period | 2.70 (2.040) | 1.52 (1.365)

5. Secondary Outcome: The Number Participants Achieving >=50% RBC Transfusion Burden Reduction From Baseline Over Any 84-Day Period (Cohorts 2 and 3B Only)
Description: The number of participants who reduce their transfusion burden by ≥ 50% from baseline over any consecutive 84-day period. Baseline is defined as average number of RBC units per 28 days over the 84 days period on or prior to the C1D1 date. The primary treatment period is from Day 1 to and including Day 168. The entire treatment period is from Day 1 through the end of treatment.
Time Frame: Baseline and from Day 1 through end of treatment (up to approximately 232 weeks).
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: RBC-Transfusion Dependent | Cohort 3B: RBC-Transfusion Dependent (Stable Dose of Ruxolitinib)
Number analyzed (Participants) | 21 | 38
Participants
  Primary Treatment Period | 10 | 19
  Entire Treatment Period | 10 | 20

6. Secondary Outcome: The Number of Participants Who Achieve ≥ 50% Reduction in Fatigue Symptom as Measured by the Myeloproliferative Neoplasms Symptom Assessment Form Total Symptom Score (MPN-SAF TSS)
Description: Symptoms response improvement will be assessed using the number of participants who achieve ≥ 50% reduction in fatigue symptoms. Fatigue is 1 out of 10 total symptoms scored on a 0 (absent/as good as it can be) to 10 (worst imaginable/as bad as it can be).
  The primary treatment period is from Day 1 to and including Day 168. The entire treatment period is from Day 1 through the end of treatment. Baseline is defined as the last value on or before the first dose of study drug.
  Last Available = Last available assessment on or before the end of the treatment period.
  Mean = Mean value of the weekly assessments over the treatment period.
Time Frame: Baseline and from Day 1 through end of treatment (up to approximately 232 weeks)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Anemia Only | Cohort 2: RBC-Transfusion Dependent | Cohort 3A: Anemia Only (Stable Dose of Ruxolitinib) | Cohort 3B: RBC-Transfusion Dependent (Stable Dose of Ruxolitinib)
Number analyzed (Participants) | 22 | 21 | 14 | 38
Participants
  Primary Treatment Period (Last Available) | 4 | 2 | 4 | 10
  Entire Treatment Period (Last Available) | 4 | 1 | 4 | 7
  Primary Treatment Period (Mean) | 5 | 1 | 3 | 5
  Entire Treatment Period (Mean) | 4 | 0 | 3 | 5

7. Secondary Outcome: The Number of Participants Who Achieve ≥ 50% Reduction in Total Symptom Score (TSS) as Measured by the Myeloproliferative Neoplasms Symptom Assessment Form Total Symptom Score (MPN-SAF TSS)
Description: TSS includes 10 items - worst fatigue, concentration, early satiety, inactivity, night sweats, itching, bone pain, abdominal discomfort, weight loss, and fevers, scored on a 0 (absent/as good as it can be) to 10 (worst imaginable/as bad as it can be). For participants who completed at least six of these 10 items, the MPN-SAF TSS was computed as the average of the observed items multiplied by 10 to achieve a 0-to-100 scale. The MPN-SAF TSS thus had a possible range of 0 to 100.
  The primary treatment period is from Day 1 to and including Day 168. The entire treatment period is from Day 1 through the end of treatment. Baseline is defined as the last value on or before the first dose of study drug.
  Last Available = Last available assessment on or before the end of the treatment period.
  Mean = Mean value of the weekly assessments over the treatment period.
Time Frame: Baseline and from Day 1 through end of treatment (up to approximately 232 weeks)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Anemia Only | Cohort 2: RBC-Transfusion Dependent | Cohort 3A: Anemia Only (Stable Dose of Ruxolitinib) | Cohort 3B: RBC-Transfusion Dependent (Stable Dose of Ruxolitinib)
Number analyzed (Participants) | 22 | 21 | 14 | 38
Participants
  Primary Treatment Period (Last Available) | 2 | 2 | 2 | 9
  Entire Treatment Period (Last Available) | 2 | 1 | 2 | 7
  Primary Treatment Period (Mean) | 2 | 2 | 3 | 6
  Entire Treatment Period (Mean) | 2 | 2 | 3 | 6

8. Secondary Outcome: Mean Changes in the Functional Assessment of Cancer Therapy - Anemia (FACT-An) Total Scores Over the Study Compared to Baseline
Description: The Functional Assessment of Cancer Therapy - Anemia (FACT-An) questionnaire includes 47 items rating on a 5-point Likert scale from 0 (not at all) to 4 (very much) on five primary subscales:
  * Physical well-being (sum of 7 items, score range from 0-28)
  * Social/Family well-being (sum of 7 items, score range from 0-28)
  * Emotional well-being (sum of 6 items, score range from 0-24)
  * Functional well-being (sum of 7 items, score range from 0-28)
  * Anemia-related symptoms (sum of 20 items, score range from 0-80)
  A total score for the FACT-An can be calculated by summing the five primary subscales with a score range from 0-188. Higher scores representing better quality of life. Baseline is defined as the last value on or before the first dose of study drug.
Time Frame: Day 169 and End of treatment (up to approximately 232 weeks)
Population: ITT population with available health related quality of life (HRQOL) assessments. (Intent-to-treat (ITT) population: All enrolled participants regardless of whether or not the participant received luspatercept.)
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1: Anemia Only | Cohort 2: RBC-Transfusion Dependent | Cohort 3A: Anemia Only (Stable Dose of Ruxolitinib) | Cohort 3B: RBC-Transfusion Dependent (Stable Dose of Ruxolitinib)
Number analyzed (Participants) | 9 | 9 | 8 | 14
Score on a scale
  Day 169: number analyzed (Participants) | 9 | 9 | 5 | 14
  Day 169 | -10.4 (13.23) | -15.7 (14.24) | -9.4 (9.24) | 5.0 (21.77)
  End of Treatment: number analyzed (Participants) | 9 | 8 | 8 | 14
  End of Treatment | -15.9 (18.35) | -16.6 (16.80) | -12.6 (10.03) | -14.2 (21.98)

9. Secondary Outcome: Mean Change in EQ-5D-5L Utility Score Compared to Baseline
Description: The European Quality of Life 5D-5L Scale (EQ-5D-5L) assesses general health-related quality of life. Health is defined in 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. Responses are coded so that a '1' indicates no problem, and '5' indicates the most serious problem. The responses for the 5 dimensions are combined in a 5-digit number. The EQ-5D-5L health utility index for this analysis will be derived using the United Kingdom (UK) value sets based on UK time trade-off (TTO) valuation techniques and will use the Decision Support Unit (DSU) model to cross-walk to the EQ-5D-3L value set from the UK to derive a single index value. The EQ-5D-3L health utility index based on the UK population weights range from -0.594 to 1.0 with higher scores indicating higher health utility.
Time Frame: Day 169 and End of treatment (up to approximately 232 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1: Anemia Only | Cohort 2: RBC-Transfusion Dependent | Cohort 3A: Anemia Only (Stable Dose of Ruxolitinib) | Cohort 3B: RBC-Transfusion Dependent (Stable Dose of Ruxolitinib)
Number analyzed (Participants) | 11 | 9 | 8 | 14
Score on a scale
  Day 169: number analyzed (Participants) | 11 | 9 | 6 | 14
  Day 169 | -0.043 (0.1466) | -0.063 (0.1152) | -0.126 (0.1246) | 0.005 (0.1084)
  End of Treatment: number analyzed (Participants) | 10 | 9 | 8 | 12
  End of Treatment | -0.029 (0.1029) | -0.120 (0.1740) | -0.129 (0.1812) | -0.103 (0.2055)

10. Secondary Outcome: The Number of Participants Treatment-Emergent Adverse Events (TEAE)
Description: TEAE is defined as any AEs that begin or worsen on or after the day of the first dose. An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. An SAE is any AE occurring at any dose that: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or constitutes an important medical event. The severity/intensity of AEs will be graded based on the Common Terminology Criteria for Adverse Events (CTCAE, version 4.03) where Grade 3 = Severe, Grade 4 = Life-threatening, and Grade 5 = Death.
Time Frame: From first dose through 42 days after the last dose (up to approximately 238 weeks)
Population: Safety population: All enrolled participants who received at least 1 dose of luspatercept.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Anemia Only | Cohort 2: RBC-Transfusion Dependent | Cohort 3A: Anemia Only (Stable Dose of Ruxolitinib) | Cohort 3B: RBC-Transfusion Dependent (Stable Dose of Ruxolitinib)
Number analyzed (Participants) | 22 | 21 | 14 | 38
Participants
  Participants with at Least One TEAE | 21 | 19 | 13 | 36
  Participants with at Least One Treatment-Related TEAE | 14 | 5 | 7 | 19
  Participants with at Least One Serious TEAE | 8 | 8 | 4 | 17
  Participants with at Least One Treatment-Related Serious TEAE | 1 | 0 | 0 | 2
  Participants with at Least One TEAE Grade >=3 | 9 | 11 | 4 | 24
  Participants with at Least One Treatment-Related TEAE Grade >=3 | 0 | 1 | 2 | 7
  Participants with at Least One TEAE Leading to Dose Interruption | 2 | 2 | 3 | 12
  Participants with at Least One Treatment-Related TEAE Leading to Dose Interruption | 1 | 1 | 1 | 4
  Participants with at Least One TEAE Leading to Dose Reduction | 1 | 0 | 2 | 2
  Participants with at Least One Treatment-Related TEAE Leading to Dose Reduction | 1 | 0 | 2 | 2
  Participants with at Least One TEAE Leading to Study Drug Withdrawn | 1 | 2 | 1 | 5
  Participants with at Least One Treatment-Related TEAE Leading to Study Drug Withdrawn | 0 | 0 | 0 | 1
  Participants with at Least One TEAE Leading to Death | 1 | 2 | 0 | 5
  Participants with at Least One Treatment-Related TEAE Leading to Death | 0 | 0 | 0 | 0

11. Secondary Outcome: CL/F (L/Day)
Description: Apparent clearance
Time Frame: C1D1 (pre-dose), C1D8, C1D15, C2D1, C4D1, C5D1, C5D8, C6D1, and C8D1, day 169, Day 1 of every 4th Extension Phase treatment cycle for up to 1 year post the date of first dose of luspatercept, and end of treatment.
Population: All treated participants with available serum concentration measurements
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/day
Arm/Group | Cohort 1: Anemia Only | Cohort 2: RBC-Transfusion Dependent | Cohort 3A: Anemia Only (Stable Dose of Ruxolitinib) | Cohort 3B: RBC-Transfusion Dependent (Stable Dose of Ruxolitinib)
Number analyzed (Participants) | 22 | 21 | 14 | 38
Liter/day | 0.61 (51) | 0.53 (31) | 0.46 (34) | 0.44 (38)

12. Secondary Outcome: V1/F (L)
Description: Apparent volume of distribution of the central compartment
Time Frame: as for outcome 11
Population: All treated participants with available serum concentration measurements
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Cohort 1: Anemia Only | Cohort 2: RBC-Transfusion Dependent | Cohort 3A: Anemia Only (Stable Dose of Ruxolitinib) | Cohort 3B: RBC-Transfusion Dependent (Stable Dose of Ruxolitinib)
Number analyzed (Participants) | 22 | 21 | 14 | 38
Liter | 11.65 (53) | 10.15 (31) | 11.36 (34) | 10.84 (39)

13. Secondary Outcome: Ka (Day-1)
Description: First-order rate constant of absorption
Time Frame: as for outcome 11
Population: All treated participants with available serum concentration measurements
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day-1
Arm/Group | Cohort 1: Anemia Only | Cohort 2: RBC-Transfusion Dependent | Cohort 3A: Anemia Only (Stable Dose of Ruxolitinib) | Cohort 3B: RBC-Transfusion Dependent (Stable Dose of Ruxolitinib)
Number analyzed (Participants) | 22 | 21 | 14 | 38
Day-1 | 0.3 (37) | 0.28 (19) | 0.29 (21) | 0.28 (28)

14. Secondary Outcome: T1/2 (Day)
Description: Elimination half-life
Time Frame: as for outcome 11
Population: All treated participants with available serum concentration measurements
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day
Arm/Group | Cohort 1: Anemia Only | Cohort 2: RBC-Transfusion Dependent | Cohort 3A: Anemia Only (Stable Dose of Ruxolitinib) | Cohort 3B: RBC-Transfusion Dependent (Stable Dose of Ruxolitinib)
Number analyzed (Participants) | 22 | 21 | 14 | 38
Day | 13.28 (2.4) | 13.3 (1.4) | 16.96 (2.1) | 16.98 (2.2)

15. Secondary Outcome: Tmax (Day)
Description: Time to reach the maximum concentration for the first dose (Cmax)
Time Frame: as for outcome 11
Population: All treated participants with available serum concentration measurements
Measure: Median (Full Range); unit: Day
Arm/Group | Cohort 1: Anemia Only | Cohort 2: RBC-Transfusion Dependent | Cohort 3A: Anemia Only (Stable Dose of Ruxolitinib) | Cohort 3B: RBC-Transfusion Dependent (Stable Dose of Ruxolitinib)
Number analyzed (Participants) | 22 | 21 | 14 | 38
Day | 6.72 [4.84 to 10.01] | 7.38 [5.75 to 9.14] | 7.85 [6.17 to 9.54] | 7.96 [5.24 to 11.34]

16. Secondary Outcome: Cmax (µg/mL)
Description: Maximum concentration for the first dose
Time Frame: as for outcome 11
Population: All treated participants with available serum concentration measurements
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Cohort 1: Anemia Only | Cohort 2: RBC-Transfusion Dependent | Cohort 3A: Anemia Only (Stable Dose of Ruxolitinib) | Cohort 3B: RBC-Transfusion Dependent (Stable Dose of Ruxolitinib)
Number analyzed (Participants) | 22 | 21 | 14 | 38
µg/mL | 4.41 (39) | 4.68 (20) | 4.96 (23) | 5.01 (30)

17. Secondary Outcome: Cmax.ss (µg/mL)
Description: Maximum concentration for the first dose (Cmax) at steady state for the starting dose
Time Frame: as for outcome 11
Population: All treated participants with available serum concentration measurements
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Cohort 1: Anemia Only | Cohort 2: RBC-Transfusion Dependent | Cohort 3A: Anemia Only (Stable Dose of Ruxolitinib) | Cohort 3B: RBC-Transfusion Dependent (Stable Dose of Ruxolitinib)
Number analyzed (Participants) | 22 | 21 | 14 | 38
µg/mL | 7.28 (42) | 7.72 (21) | 9.45 (24) | 9.6 (32)

18. Secondary Outcome: AUCss (Day* µg/mL)
Description: Area under the concentration-time curve at the steady state for the starting dose
Time Frame: as for outcome 11
Population: All treated participants with available serum concentration measurements
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day* µg/mL
Arm/Group | Cohort 1: Anemia Only | Cohort 2: RBC-Transfusion Dependent | Cohort 3A: Anemia Only (Stable Dose of Ruxolitinib) | Cohort 3B: RBC-Transfusion Dependent (Stable Dose of Ruxolitinib)
Number analyzed (Participants) | 22 | 21 | 14 | 38
day* µg/mL | 123 (47) | 132 (24) | 168 (26) | 171 (35)

19. Secondary Outcome: The Number of Participants With Antidrug Antibody (ADA) Measurements
Description: The ADA status of a participant during treatment is determined based on the longitudinal ADA results as follows:
  Negative: All samples (baseline and post-baseline) are negative. Positive to treatment-emergent ADA: At least one post-baseline sample is positive if the baseline sample is negative, or at least one post-baseline sample is positive with a titer ≥ 4-fold of the baseline titer if the baseline sample is positive
Time Frame: C1D1 (pre- dose), C2D1, C4D1, C6D1, C8D1, Day 1 of every 4th Extension Phase treatment cycle for up to 1 year post the date of first dose of luspatercept, and end of treatment.
Population: Safety population: All enrolled participants who received at least 1 dose of luspatercept.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Anemia Only | Cohort 2: RBC-Transfusion Dependent | Cohort 3A: Anemia Only (Stable Dose of Ruxolitinib) | Cohort 3B: RBC-Transfusion Dependent (Stable Dose of Ruxolitinib)
Number analyzed (Participants) | 22 | 21 | 14 | 38
Participants
  Positive | 1 | 2 | 2 | 2
  Negative | 21 | 19 | 12 | 36

20. Secondary Outcome: Mean Changes in Hemoglobin Over the Study Compared to Baseline in the Absence of RBC Transfusions (Cohorts 1 and 3A)
Description: Calculated based on average hemoglobin measurements collected during the treatment period.The primary treatment period is from Day 1 to and including Day 168. The entire treatment period is from Day 1 through the end of treatment. The baseline RBC transfusion is defined as average number of RBC units/28 days over the 84 days period immediately prior to the C1D1 date.
Time Frame: Baseline and Day 1 through end of treatment (up to approximately 232 weeks)
Population: Intent-to-treat (ITT) population: All enrolled participants regardless of whether or not the participant received luspatercept. Pre-specified to be collected for Cohorts 1 and 3A only.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Cohort 1: Anemia Only | Cohort 3A: Anemia Only (Stable Dose of Ruxolitinib)
Number analyzed (Participants) | 22 | 14
g/dL
  Primary Treatment Period | 0.795 (0.7697) | 1.157 (0.5178)
  Entire Treatment Period | 0.824 (0.8613) | 1.172 (0.5992)

21. Secondary Outcome: The Number of Participants With a Mean Hemoglobin Increase >= 1.5 g/dL From Baseline Over Any Consecutive 84-day Period (Cohorts 1 and 3A)
Description: The number of participants with a Mean hemoglobin increase of ≥ 1.5 g/dL from baseline over any consecutive 84-day period without an RBC transfusion. The primary treatment period is from Day 1 to and including Day 168. The entire treatment period is from Day 1 through the end of treatment. Baseline is defined as all non-missing Hgb records within 28 days on or prior to date of first dose (or date of enrollment if not treated).
Time Frame: Baseline and Day 1 through end of treatment (up to approximately 232 weeks)
Population: Intent-to-treat (ITT) population: All enrolled participants regardless of whether or not the participant received luspatercept. Prespecified to be reported for Cohorts 1 and 3A only.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Anemia Only | Cohort 3A: Anemia Only (Stable Dose of Ruxolitinib)
Number analyzed (Participants) | 22 | 14
Participants
  Primary Treatment Period | 5 | 6
  Entire Treatment Period | 6 | 7

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their first dose to their study completion (up to approximately 4 years and 8 months) SAEs and Other AEs were assessed from first dose through 42 days after the last dose (up to approximately 238 weeks)
Arm/Group | Cohort 1: Anemia Only | Cohort 2: RBC-Transfusion Dependent | Cohort 3A: Anemia Only (Stable Dose of Ruxolitinib) | Cohort 3B: RBC-Transfusion Dependent (Stable Dose of Ruxolitinib)
All-Cause Mortality (participants affected / at risk) | 6/22 | 12/21 | 2/14 | 13/38
Serious Adverse Events (participants affected / at risk) | 8/22 | 8/21 | 4/14 | 17/38
Other Adverse Events (participants affected / at risk) | 21/22 | 19/21 | 13/14 | 33/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Anemia Only (N=22) | Cohort 2: RBC-Transfusion Dependent (N=21) | Cohort 3A: Anemia Only (Stable Dose of Ruxolitinib) (N=14) | Cohort 3B: RBC-Transfusion Dependent (Stable Dose of Ruxolitinib) (N=38)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0
Gait disturbance (General disorders) | 1 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Biliary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Cerebral toxoplasmosis (Infections and infestations) | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 1 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 1
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 1 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 1
Troponin T increased (Investigations) | 0 | 0 | 0 | 1
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 2
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Skin squamous cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 2 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Aortic embolus (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Anemia Only (N=22) | Cohort 2: RBC-Transfusion Dependent (N=21) | Cohort 3A: Anemia Only (Stable Dose of Ruxolitinib) (N=14) | Cohort 3B: RBC-Transfusion Dependent (Stable Dose of Ruxolitinib) (N=38)
Anaemia (Blood and lymphatic system disorders) | 3 | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 2
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 3 | 1 | 11
Hypothyroidism (Endocrine disorders) | 2 | 0 | 0 | 2
Glaucoma (Eye disorders) | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 5 | 2 | 2 | 4
Constipation (Gastrointestinal disorders) | 2 | 2 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 4 | 4 | 11
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 3 | 2 | 6
Vomiting (Gastrointestinal disorders) | 2 | 0 | 2 | 2
Asthenia (General disorders) | 1 | 3 | 0 | 5
Chills (General disorders) | 0 | 1 | 1 | 1
Early satiety (General disorders) | 0 | 0 | 2 | 2
Fatigue (General disorders) | 4 | 5 | 2 | 6
Influenza like illness (General disorders) | 1 | 1 | 3 | 1
Injection site pain (General disorders) | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 2 | 0 | 0 | 1
Oedema peripheral (General disorders) | 3 | 0 | 1 | 5
Pain (General disorders) | 0 | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 1 | 1 | 0
Pyrexia (General disorders) | 5 | 1 | 1 | 7
Abscess limb (Infections and infestations) | 0 | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 2
Cystitis (Infections and infestations) | 1 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 2
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 1 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 2 | 2
Urinary tract infection (Infections and infestations) | 2 | 4 | 1 | 3
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 4
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 1 | 3
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 1 | 7
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 2 | 0
Blood glucose increased (Investigations) | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 2 | 0 | 1
White blood cell count increased (Investigations) | 0 | 0 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0 | 2
Gout (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 3
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 3 | 4
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 4
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 3
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Disturbance in attention (Nervous system disorders) | 0 | 0 | 1 | 2
Dizziness (Nervous system disorders) | 2 | 2 | 3 | 7
Headache (Nervous system disorders) | 3 | 1 | 1 | 3
Memory impairment (Nervous system disorders) | 0 | 1 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 2
Depression (Psychiatric disorders) | 2 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 2 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 3
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 0 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 2 | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 2 | 3 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2 | 3 | 3
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 5 | 3 | 6 | 9
Hypotension (Vascular disorders) | 0 | 0 | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-19): https://cdn.clinicaltrials.gov/large-docs/42/NCT03194542/Prot_SAP_000.pdf